CLINICAL TRIAL: NCT01007279
Title: ROsuvastatin Pretreatment in Patients Undergoing Elective PCI to Reduce the Incidence of MyocArdial Periprocedural Necrosis
Brief Title: Rosuvastatin in Preventing Myonecrosis in Elective Percutaneous Coronary Interventions (PCIs)
Acronym: ROMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: GENNARO SARDELLA, POLICLINICO UMBERTO I-SAPIENZA UNIVERSITY OF ROME
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMA55
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-03

CONDITIONS: Periprocedural Myocardial Necrosis
Keywords: Percutaneous angioplasty; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLOPIDOGREL (Active Comparator)
  Interventions: Drug: ROSUVASTATIN
- ROSUVASTATIN (Experimental)
  Interventions: Drug: ROSUVASTATIN

INTERVENTIONS:
Drug: ROSUVASTATIN — 40 mg before procedure

SUMMARY:
An increase in cardiac biomarkers has been shown to occur in 5% to 30% of patients after otherwise successful percutaneous coronary interventions (PCIs)(1) Apart from side-branch occlusion, intimal dissection and coronary spasm, a possible aetiology of myonecrosis after PCI might be distal embolization of atherogenic materials from plaque disruption,(2 )causing obstruction of blood flow at capillary level resulting in micro-infarction.(3,4 )Recent studies have suggested that pretreatment with Atorvastatin may be associated with a reduction in infarct size after elective PCI. (5-7 ).Actually the standard pretreatment in patients undergoing elective coronary-PCI and already treated with aspirin is copidogrel loading dose administration before procedure.(8,9 ) The investigators hypothesized that a high (40mg) loading dose of Rosuvastatin administered within 24h before the procedure may be effective in reducing the rate of periprocedural MI.Therefore, the investigators will conduct a single center,prospective randomized study to assess whether a single,high (40mg) loading (within24h)dose of Rosuvastatin is effective in preventing elevation of biomarkers of MI after elective coronary stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina

Exclusion Criteria:

* Baseline myocardial enzyme rise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Myocardial enzymes arise | 6-12-24 hours

SECONDARY OUTCOMES:
MACE | 1-6-9 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I, Rome, Italy